CLINICAL TRIAL: NCT05640869
Title: The Diabetes Prevention Program to Treat Overweight and Obesity
Brief Title: Diabetes Prevention Program to Treat Overweight and Obesity
Acronym: DPP-TOO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Courtney E Gamston, Professor of Experiential Practice, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-254 EP 2207
Record Dates: First submitted 2022-08-22; First posted 2022-12-07 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Weight Loss; PreDiabetes
Keywords: community pharmacy
MeSH Terms: conditions — Weight Loss; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified DPP (Experimental): Participants in this arm will participate in the modified Diabetes Prevention Program curriculum.
  Interventions: Behavioral: Modified Diabetes Prevention Program Curriculum

INTERVENTIONS:
Behavioral: Modified Diabetes Prevention Program Curriculum — The modified DPP curriculum will be an exact copy of the current DPP curriculum except that references to the prevention of diabetes will be modified to prevention of health outcomes associated with overweight/obesity and/or management of overweight/obesity.

SUMMARY:
The purpose of this study is to demonstrate the efficacy of the diabetes prevention program for the treatment of overweight and obesity within the community pharmacy setting. The long-term goal is to demonstrate the potential to improve diabetes prevention efforts through expanded access to weight loss services provided in community pharmacies.

DETAILED DESCRIPTION:
An estimated 38% percent of U.S. adults currently has prediabetes. In individuals aged 65 years and older, the prevalence of prediabetes is 48.8%. Prediabetes is commonly a precursor to the development of type 2 diabetes (t2d). Approximately 5-10% of individuals with prediabetes progress to t2d annually, with 70% developing t2d within their lifetime. Obesity is a significant risk factor for both prediabetes and diabetes, and its prevalence is steadily increasing. In 2020, a combined 66.7% of U.S. adults were classified as overweight or obese. In individuals with prediabetes, interventions leading to a 5-10% decrease in baseline body weight decrease the risk for progression to t2d by 58% at three years and 71% for those aged 60 years and older. At ten and fifteen years, the risk was decreased by 34% and 27%, respectively, and diabetes progression was significantly delayed. Based on these findings, a structured lifestyle intervention program was developed and has been available for public use by the Centers for Disease Control and Prevention (CDC) since 2010. Despite significant resources for the implementation of the Diabetes Prevention Program (DPP), program dissemination and utilization remains low. There are currently 1,882 registered DPP providers nationwide. Due to the modest results attributed to significant efforts to increase the access to and participation in DPP programs across the country, consideration should be given to modifying the current approach to diabetes prevention efforts.

In 2020, approximately 42.4% of American adults had obesity according to the 2021 State of Obesity: Better Policies for a Healthier America report. The prevalence of obesity has been steadily increasing for the last two decades. This upward trend is expected to continue this if effective and sustainable solutions are not employed. According to the CDC, in 2013-2016, 49.1% of adults reported having tried to lose weight within the last year. Searching "weight loss" in any internet browser will return over a billion results ranging from diet plans and weight loss programs to testimonials of individual weight loss journeys. Due to the prevalence of overweight and obesity, the demand for weight loss interventions, and the efficacy of weight reduction for decreasing the risk for t2d development, expanding access to evidence-based weight loss interventions has the potential to significantly advance diabetes prevention efforts nationwide by shifting the focus from preventing prediabetes to treating overweight and obesity. One major gap in the current treatment landscape is how to implement an effective program for adult weight loss with widespread impact.

Given the prevalence and visibility of community pharmacies, this setting is ideal for the dissemination of weight management services. In order to assess the potential impact, this pilot study aims to implement a modified-DPP program and to assess the diabetes risk and health outcomes of individuals choosing to participate in the program..

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* BMI ≥ 25kg/m2 (23 if Asian)

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 6 months
  Change from baseline body weight
Change in A1c | 3- and 6- months
  Change from baseline A1c

SECONDARY OUTCOMES:
Proportion of patients meeting DPP program criteria | From enrollment, assessed once enrollment is complete, within 3 months of study start.
  Percentage of individuals meeting DPP criteria at baseline
Blood pressure change | 6 months
  Change from baseline blood pressure
Physical activity change | 6 months
  Change from baseline self-reported physical activity in minutes per week

OTHER OUTCOMES:
Participation and attrition | 6 months
  Rate of participation and attrition
Reasons for participation/non-participation | 1 year
  Qualitative analysis through semi-structured interview
Change in level of confidence in ability to motivate oneself to maintain dietary and physical activity behaviors for at least 6 months | 6 months
  Change from baseline in level of confidence in motivating oneself to engage the included dietary and physical behaviors for at lease six months as assessed by "Self-efficacy for diet and exercise behaviors" tool. Domains include sticking to an exercise regimen, making time for exercise, sticking to a diet, reducing calories, reducing salt, and reducing fat. Scale 1 to 5; higher = more confident
Change in Stage of Change for Weight Loss | 6 months
  Change from baseline in stage of change (scale 1-5; 1= precontemplation, 2= contemplation, 3= preparation, 4= action, 5= maintenance)
Change in Processes of Change for Weight Loss including the following processes: emotional re-evaluation, weight consequences evaluation, supporting relationships, and weight management actions | 6 months
  Change from baseline in process of change (scale 0 to 100; higher = more active use of the process of change)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney E Gamston, PharmD, Principal Investigator — Auburn University Harrison School of Pharmacy
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tabak AG, Herder C, Rathmann W, Brunner EJ, Kivimaki M. Prediabetes: a high-risk state for diabetes development. Lancet. 2012 Jun 16;379(9833):2279-90. doi: 10.1016/S0140-6736(12)60283-9. Epub 2012 Jun 9. PMID 22683128
- [Background] Venkataramani M, Pollack CE, Yeh HC, Maruthur NM. Prevalence and Correlates of Diabetes Prevention Program Referral and Participation. Am J Prev Med. 2019 Mar;56(3):452-457. doi: 10.1016/j.amepre.2018.10.005. Epub 2019 Jan 17. PMID 30661888
- [Background] Joiner KL, McEwen LN, Hurst TE, Adams MP, Herman WH. Domains from the health belief model predict enrollment in the National Diabetes Prevention Program among insured adults with prediabetes. J Diabetes Complications. 2022 Jul;36(7):108220. doi: 10.1016/j.jdiacomp.2022.108220. Epub 2022 May 17. PMID 35613987
- [Background] Martin CB, Herrick KA, Sarafrazi N, Ogden CL. Attempts to Lose Weight Among Adults in the United States, 2013-2016. NCHS Data Brief. 2018 Jul;(313):1-8. PMID 30044214
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Andres A, Saldana C, Gomez-Benito J. Establishing the stages and processes of change for weight loss by consensus of experts. Obesity (Silver Spring). 2009 Sep;17(9):1717-23. doi: 10.1038/oby.2009.100. Epub 2009 Apr 9. PMID 19360014
- See also: CDC Nutrition, Physical Activity, and Obesity: Data, Trends and Maps — https://www.cdc.gov/nccdphp/dnpao/data-trends-maps/index.html
- See also: NIH Diabetes Prevention Program — https://www.niddk.nih.gov/about-niddk/research-areas/diabetes/diabetes-prevention-program-dpp
- See also: Prediabetes Risk Test — https://www.cdc.gov/prediabetes/pdf/Prediabetes-Risk-Test-Final.pdf